CLINICAL TRIAL: NCT02289365
Title: Phase 2 Study of Orally Administrated JBM-TC4 for the Prevention of Acute Radiation-induced Dermatitis in Breast Cancer Patients
Brief Title: Orally Administrated JBM-TC4 Prevents Acute Radiodermatitis in Breast Cancer Patients
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Joben Bio-Medical Co., Ltd. (Industry)
Collaborators: Kaohsiung Medical University Chung-Ho Memorial Hospital (Other); Taipei Veterans General Hospital, Taiwan (Other Government); Efficient Pharma Management Corp. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: JBM-001; IND 117691 (Other: U.S. Food and Drug Administration)
Record Dates: First submitted 2014-11-05; First posted 2014-11-13 (Estimated); Last update posted 2016-06-15 (Estimated); Status verified 2016-06

CONDITIONS: Radiodermatitis
Keywords: Radiodermatitis; Breast cancer; Radiotherapy
MeSH Terms: conditions — Radiodermatitis; Breast Neoplasms

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Group I (Placebo Comparator): Totally 3000 mg of PEG-400 per day. 3 capsules of 500 mg PEG-400 per time, twice a day.
  Interventions: Drug: 3000 mg of PEG-400 per day
- Group II (Experimental): Totally 2000 mg of JBM-TC4 per day. 2 capsules of 500 mg JBM-TC4 plus 1 capsule of 500 mg PEG-400 per time, twice a day.
  Interventions: Drug: 2000 mg of JBM-TC4 per day
- Group III (Experimental): Totally 3000 mg of JBM-TC4 per day. 3 capsules of 500 mg JBM-TC4 per time, twice a day.
  Interventions: Drug: 3000 mg of JBM-TC4 per day

INTERVENTIONS:
Drug: 2000 mg of JBM-TC4 per day — 2 capsules of 500 mg JBM-TC4 plus 1 capsule of 500 mg PEG-400, oral route per time twice a day in Day (-7) prior to radiotherapy and continue through the radiotherapy period for additional 11 weeks.
  Arms: Group II
Drug: 3000 mg of JBM-TC4 per day — 3 capsules of 500 mg JBM-TC4, oral route per time twice a day in Day (-7) prior to radiotherapy and continue through the radiotherapy period for additional 11 weeks.
  Arms: Group III
Drug: 3000 mg of PEG-400 per day — 3 capsules of 500 mg polyethylene glycol 400 (PEG-400), oral route per time twice a day in Day (-7) prior to radiotherapy and continue through the radiotherapy period for additional 11 weeks.
  Arms: Group I

SUMMARY:
This trial is designed as a multicenter, double-blinded, randomized, placebo controlled study to assess the safety and efficacy of JBM-TC4 for the prevention and treatment of acute radiation-induced dermatitis in breast cancer patients receiving radiotherapy.

DETAILED DESCRIPTION:
This study will be conducted in 2 sites in Taiwan. Upon confirmation of meeting all eligibility criteria, will be randomized in a 1:1:1 ratio to 2000 mg or 3000 mg JBM-TC4 oral treatment group or to placebo control group.

The treatment will start one week prior to radiotherapy and continue through the radiotherapy period for additional 11 weeks of JBM-TC4. The patients will take 3 treatment capsules twice a day, after breakfast and dinner. Screening visit will occur up to 14 days prior to randomization (Day 0), and informed consent form will be signed and patient eligibility criteria will be verified.Medical history information, chemistry/hematology evaluation, serum pregnancy will be conducted and documented. On Day 0, baseline assessment will be done and study drug will be dispensed. The patients will be instructed to start their study medication after breakfast on Day 1 and record the administration time in the study diary. Post-operative radiotherapy will begin for all patients after taking the treatment for 7 days. On Days 8, 15, 22, 29, 36, 43, 50, 57, 64, 71, 78, 85 and 92, data including radiation dermatitis severity, redness and pain scale will be collected when patients return to the clinic for evaluation. On Days 29, 57, 85 and 92, quality of life questionnaire will be completed by patients and blood will be drawn for chemistry/hematology evaluation. The final study visit will occur one week after the last dose of study medication, which will be around Day 92. ECG will be evaluated on Day 8 and 92. A total of 120 women with breast cancer will be recruited into this study. Safety will be assessed through recording of adverse events, assessment of vital signs, and chemistry/hematology laboratory testing. During each clinic visit, investigator will take down the vital signs of the patients and ask if the patients has experienced any adverse events. All information will be recorded on the case report form.

The primary efficacy endpoint in this study is to assess the effectiveness of JBM-TC4 for the prevention and treatment of acute radiation-induced dermatitis. The effectiveness will be determined by the recording of the radiation dermatitis severity scale for patients during each weekly study visit. Secondary efficacy endpoint include 1) Presence of moist desquamation and 2) redness at the radiation treated site at any visit. 3)The worst pain related to dermatitis between baseline and follow-up visit at the radiotherapy site. 4) Quality of life and 5) safety evaluation assessment. At the final visit, each investigator will be ask to rate their patients' responses to treatment.

ELIGIBILITY:
Inclusion Criteria:

* males or non-pregnant females at least 20 year of age.
* Diagnosis of, non-inflammatory breast adenocarcinoma and be referred for post-operative radiotherapy without concurrent chemotherapy.
* Breast adenocarcinoma previously treated by lumpectomy with or without adjuvant or neoadjuvant chemotherapy or hormonal treatment.
* With in situ breast cancer are also eligible
* Prescribed concurrent hormone treatment with radiation treatment
* Participants must be scheduled to receive 5 sessions of radiotherapy per week (1 session per day) for at least 5 weeks using standard (1.8 Gy to 2.0 Gy per session) for total dose of at least 45 Gy.
* A time period of 3 weeks must elapse after chemotherapy and surgery before beginning this study.
* Must be able to swallow medication.
* Participant must give informed consent.

Exclusion Criteria:

* Bilateral breast cancer
* Previous radiotherapy to the breast or chest.
* Chemotherapy cocurrent with radiation treatment.
* Receiving treatment with anti-coagulants, or anti-human epidermal growth factor receptor drugs, e.g., Iressa (gefitinib), Erbitux (cetuximab, C225), concurrently with their radiotherapy.
* Prior breast reconstructions, implants, and/or expanders.
* Known radiosensitivity syndromes, e.g., Ataxia-telangiectasia.
* Collagen vascular disease, vasculitis, unhealed surgical sites, breast infections, or systemic lupus erythematosus.
* Baseline blood tests that meet the following criteria:

  * Grade 2 change in hemoglobin (i.e., 25% decease from baseline);
  * Grade 1 change in platelets (i.e., < 75'000/mm3);
  * Grade 2 change in prothrombin time and partial thromboplastin time (i.e., 1.5-2x upper limit of normal);
  * Grade 1 change in aspartate transaminase, alanine transaminase (i.e., > 2.5x upper limit of normal);
  * Grade 1 change in bilirubin (i.e., > 1.5x upper limit of normal);
  * Grade 1 change in Creatinine (i.e., > 2x upper limit of normal).
* Conditions affecting the absorption for oral medications.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2014-11; Primary Completion 2016-12 (Estimated); Study Completion 2016-12 (Estimated)

PRIMARY OUTCOMES:
Radiation Dermatitis Severity Scale (RDS) | baseline to 92 days
  During each weekly visit (Day 0,8, 15, 22, 29, 36, 43, 50, 57, 64, 71, 78, 86 and 92), starting from baseline evaluation at Day 0, the severity of radiodermatitis in breast cancer patients at the radiotherapy site will be assess by the investigator using the RDS (CTCAE 4.03), which the ranges from 0 to 5 with increments of 1.

SECONDARY OUTCOMES:
Presence of Moist Desquamation | baseline to 92 days
  The presence of moist desquamation information will be obtained from RDS score at 0,8, 15, 22, 29, 36, 43, 50, 57, 64, 71, 78, 86, 92 days. Patients with score 3 or more will be recorded as having moist desquamation on the radiotherapy site.
Redness Scale | baseline to 92 days
  Score of redness at the radiotherapy site will be evaluated at all the visits starting from Day 0 along with RDS scale (at 0,8, 15, 22, 29, 36, 43, 50, 57, 64, 71, 78, 86, 92 days).
Worst Pain Related to Radiodermatitis at the site | baseline to 92 days
  Starting on Day 0, patients will be ask to circle a number that best describe the worst pain related to dermatitis they have been experiencing through the past week. (at 0,8, 15, 22, 29, 36, 43, 50, 57, 64, 71, 78, 86, 92 days)
Improve Quality of Life | 92 days
  Quality of life is measured using the Quality of Life Questionnaire. Patients will select the response that best describe their conditions at Day 0, 29, 57, 85 and 92. Scores will be calculated ans transcribed scores will be collected on the case report forms.
Vital sign | baseline to 92 days
  Blood pressure and pulse rate will be measured in the writing arm and recorded to mmHg or beat per minute, respectively. The same arm will be used through this study. They will be measured after 5 minutes supine and 2 minutes standing. Oral temperature, recorded to the nearest 0.1 degree Celsius, will be measured during the supine vital sign measurements. All above will be obtained at Day 0,8, 15, 22, 29, 36, 43, 50, 57, 64, 71, 78, 86 and 92.
Electrocardiogram | baseline to 85 days
  A 12-lead ECG will be obtained on all subjects at the designed times (Fay 0, 8, 29, 57 and 85) in the flow charts.
Hematology and Serology test | baseline to 92 days
  During the visits on Days 0, 29, 57, 85 and 92, the blood samples will be drawn for routine laboratory evaluations. The parameters includes hemoglobin, hematocrit, white blood count with differential, platelet count, red blood cell count, Glutamate-oxaloacetate transaminase, Glutamic-Pyruvic Transaminase, blood urea nitrogen, creatinine, cholesterol, HDL, LDL, triglyceride, blood glucose test.. Plasma sample will be collected and frozen at visits days 0, 8 (after ECG collection), 29, 57 and 85 for future assay of pharmacokinetics.
Occurrence of Adverse Events | up to 92 days
  All adverse events, regardless of seriousness, severity, or presumed relationship to study drug, are events that occur between the day of with the informed consent is signed and completion of the treatment phase. They must be recorded using medical terminology in the source document and the Case Report Form. Graphical techniques may also be used to examine the relationship between these measures and dose and to investigate any trends in the data. Incidence rates for all adverse events , and the number of subjects withdrawing from the study for each reason will be tabulated.

CONTACTS AND LOCATIONS:
Overall Officials: Chih-Jen Huang, MD-PhD, Principal Investigator — Kaohsiung Medical University Chung-Ho Memorial Hospital; Cheng-Ying Shiau, MD, Principal Investigator — Taipei Verterans General Hospital; Chin-Nan Chu, MD, Principal Investigator — China Medical University Hospital
Locations (3):
- Taiwan (3):
  - Departmant of Radiotherapy, Kaohsiung Medical University Chung-Ho Memorial Hospital, Kaohsiung, Taiwan
  - Department of Oncology, Taipei Verterans General Hospital, Taipei, Taiwan
  - Department of Radiation Oncology, China Medical University Hospital, Taichung

REFERENCES:
- [Background] Chang HC, Huang YC, Hung WC. Antiproliferative and chemopreventive effects of adlay seed on lung cancer in vitro and in vivo. J Agric Food Chem. 2003 Jun 4;51(12):3656-60. doi: 10.1021/jf021142a. PMID 12769541
- [Background] Chen HJ, Lo YC, Chiang W. Inhibitory effects of adlay bran (Coix lachryma-jobi L. var. ma-yuen Stapf) on chemical mediator release and cytokine production in rat basophilic leukemia cells. J Ethnopharmacol. 2012 May 7;141(1):119-27. doi: 10.1016/j.jep.2012.02.009. Epub 2012 Feb 14. PMID 22353428
- [Background] Chung CP, Hsu CY, Lin JH, Kuo YH, Chiang W, Lin YL. Antiproliferative lactams and spiroenone from adlay bran in human breast cancer cell lines. J Agric Food Chem. 2011 Feb 23;59(4):1185-94. doi: 10.1021/jf104088x. Epub 2011 Feb 1. PMID 21284381
- [Background] Chung CP, Hsia SM, Lee MY, Chen HJ, Cheng F, Chan LC, Kuo YH, Lin YL, Chiang W. Gastroprotective activities of adlay (Coix lachryma-jobi L. var. ma-yuen Stapf) on the growth of the stomach cancer AGS cell line and indomethacin-induced gastric ulcers. J Agric Food Chem. 2011 Jun 8;59(11):6025-33. doi: 10.1021/jf2009556. Epub 2011 May 5. PMID 21517098
- [Background] Hung WC, Chang HC. Methanolic extract of adlay seed suppresses COX-2 expression of human lung cancer cells via inhibition of gene transcription. J Agric Food Chem. 2003 Dec 3;51(25):7333-7. doi: 10.1021/jf0340512. PMID 14640580
- [Background] Kuo CC, Shih MC, Kuo YH, Chiang W. Antagonism of free-radical-induced damage of adlay seed and its antiproliferative effect in human histolytic lymphoma U937 monocytic cells. J Agric Food Chem. 2001 Mar;49(3):1564-70. doi: 10.1021/jf001215v. PMID 11312897
- [Background] Kuo CC, Chen HH, Chiang W. Adlay ( yi yi; "soft-shelled job's tears"; the seeds of Coix lachryma-jobi L. var. ma-yuen Stapf) is a Potential Cancer Chemopreventive Agent toward Multistage Carcinogenesis Processes. J Tradit Complement Med. 2012 Oct;2(4):267-75. doi: 10.1016/s2225-4110(16)30112-2. PMID 24716141
- [Background] Lee MY, Lin HY, Cheng F, Chiang W, Kuo YH. Isolation and characterization of new lactam compounds that inhibit lung and colon cancer cells from adlay (Coix lachryma-jobi L. var. ma-yuen Stapf) bran. Food Chem Toxicol. 2008 Jun;46(6):1933-9. doi: 10.1016/j.fct.2008.01.033. Epub 2008 Feb 12. PMID 18331775
- [Background] Li SC, Chen CM, Lin SH, Chiang W, Shih CK. Effects of adlay bran and its ethanolic extract and residue on preneoplastic lesions of the colon in rats. J Sci Food Agric. 2011 Feb;91(3):547-52. doi: 10.1002/jsfa.4219. Epub 2010 Nov 19. PMID 21218491
- [Background] Yao HT, Lin JH, Chiang MT, Chiang W, Luo MN, Lii CK. Suppressive effect of the ethanolic extract of adlay bran on cytochrome P-450 enzymes in rat liver and lungs. J Agric Food Chem. 2011 Apr 27;59(8):4306-14. doi: 10.1021/jf200117m. Epub 2011 Mar 18. PMID 21395288
- [Background] Zhan YP, Huang XE, Cao J, Lu YY, Wu XY, Liu J, Xu X, Xiang J, Ye LH. Clinical safety and efficacy of Kanglaite(R) (Coix Seed Oil) injection combined with chemotherapy in treating patients with gastric cancer. Asian Pac J Cancer Prev. 2012;13(10):5319-21. doi: 10.7314/apjcp.2012.13.10.5319. PMID 23244156